CLINICAL TRIAL: NCT04716543
Title: One-health Approach in Epidemiological Investigation of SARS-CoV-2 in Laos
Brief Title: Epidemiological Investigation of COVID-19 in Laos Using a One-Health Approach in Human and Animals
Acronym: LACOVISS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Centre d'Infectiologie Charles Mérieux (Other); University Hospital, Caen (Other); Department of livestock and fisheries National animal health laboratory, Vientiane, Laos (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANRS COV20 LACOVISS
Record Dates: First submitted 2020-12-14; First posted 2021-01-20 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Influenza -Like Illness; Covid19
Keywords: SARS-CoV-2; Lao PDR; One Health; virus; coronavirus; reservoir; animal; antibody; serology; PCR
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and saliva swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ILI Investigation: The suspected ILI cases will be first identified using the WHO clinical case definition of ILI and Covid 19 as either with:Acute onset of fever (> 37.5˚C axillary temperature or > 38˚C tympanic temperature) AND cough; OR Acute onset of ANY ONE OR MORE of the following signs or symptoms: Fever, cough, general weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnoea, anosmia (loss of smell) or ageusia (loss of taste); with symptoms with onset within the last 10 days.
  Interventions: Diagnostic Test: ILI and COVID-19 detection

INTERVENTIONS:
Diagnostic Test: ILI and COVID-19 detection — All participants presenting with ILI symptoms will have non-invasive exam for SARS-CoV-2 detection (nasal, throat, swab, saliva) and a questionnaire.
  All family members more than 6 months living with SARS-CoV-2 positive individuals will have will have non-invasive exam for SARS-CoV-2 detection (nasal, throat, swab, saliva) and a questionnaire.

SUMMARY:
The Respiratory infection COVID-19, due to a new coronavirus, SARS-CoV2, appeared in December 2019 in several people who attended the wildlife market in Wuhan, Hubei Province, China. While COVID-19 has spread to nearly 200 countries and caused two millions infections, Lao PDR detected its first confirmed case very recently, on March 20, three months after the start of the outbreak in China. As of April 12th, 2020, Lao PDR has only recorded 18 confirmed cases, a very low number compared to other countries around the world.

However, several key factors suggest that Lao PDR could be much more affected by COVID-19 because of the following reasons: (i) The multiple and massive trans-border movements between Lao PDR and China. (ii) The similar biogeographical and socio-ecological characteristics with South-Western China. (iii) The detection of a high diversity of Betacoronavirus sequences in several species of bats in Lao PDR. (iv) The numerous markets selling high volumes of local wildlife including bats and pangolins.

LACOVISS project aim at investigating, using a ONE-HEALTH approach, this unexpected epidemiological pattern of SARS-CoV-2 in Lao PDR by bringing together an interdisciplinary team of experts in the field from IRD, the University of Caen, the Center of Infectiology Lao-Christophe Mérieux (CILM) and the National animal Health Laboratory (NAHL) in Vientiane. The study will focus on a community-based cohort of 1092 households, including 5400 study participants, followed-up between March 2015 and February 2019 for influenza-like illness investigation and causative agents detection (LACORIS project), located in the Vientiane metropolitan area. The COVID-19 progression in Lao PDR, and track SARS-CoV-2, will be followed retrospectively and prospectively, in all potential actors in SARS-CoV-2 circulation, including humans, domestic animals, and wildlife.

The LACOVISS project will undoubtedly bring new insight in SARS-Cov-2 and SARS-CoV-like circulation in Lao PDR as well as valuable information on the natural history of COVID-19, and on the modalities of the spillover into humans, which are still largely unknown.

DETAILED DESCRIPTION:
1. INTRODUCTION

   This project is mainly based on two major questions that remain unsolved. The first one is the origin of the outbreak and the events that led to the transmission of SARS-CoV-2 to humans. The second is the striking epidemiological situation in Laos, in which only a few cases have been observed despite similar biogeographical and socio-ecological characteristics shared with South-Western China.The diversity of wild fauna (notably in southern China and in South-East Asia, where bat diversity peaks to over 100 species), associated with the wide circulation of coronaviruses, especially in Laos PDR, and their evolutionary and zoonotic potential, indicate that (past or future) emergences in Laos can be expected. In addition, given the massive population movement between Laos and China, it was expected a significant spread of COVID-19 from China to Laos. In order to respond to these two main questions, the investigators formulate the following working hypotheses to address in this project.

   Assumption 1: COVID-19 may massively spread to the Laos population in the near future through the arrival in the country of infected individuals.

   Assumption 2: SARS-CoV-2 has been already circulating in Laos before the appearance of COVID-19 outbreak in China.

   Assumption 3: SARS-CoV-2 may jump from wildlife and emerge into the Lao human population in the future Assumption 4: Some genetic closely related viruses (SARS-CoV-2-like viruses) have already circulated in Laos.
2. OBJECTIVES

   The general objective of the project is to elucidate the natural history of COVID-19 by investigating the circulation of the virus in Lao PDR following a ONE-HEALTH approach before (retrospective approach) and after (prospective approach) the initial appearance of the outbreak in China.

   In particular, the investigators will investigate the progressions of the outbreak and the reasons behind the relative low number of COVID-19 positive patients observed to date in the country, despite sharing biogeographical and socio-ecological features and trans-border with South-Western China.

   Under this general heading, the secondary objectives are:

   In humans:

   To determine COVID-19 circulation within the cohort before the appearance of the first positive cases in December 2019 in Wuhan, China To determine COVID-19 progression, over a one-year period from the beginning of the project To evaluate the SARS-CoV-2 asymptomatic infections To assess past SARS-CoV-2 circulation

   In animals:

   To investigate SARS-CoV-2 transmission to pets and domestic animals
3. METHODOLOGY

   In humans:

   The project will be conducted within a community-based cohort of 1092 households, including 5400 study participants, followed-up between March 2015 and February 2019 for influenza-like illness investigation and causative agents detection (LACORIS project, Respiratory Infectious Disease among Cohorts in Vientiane Capital, Lao PDR), located in the Vientiane metropolitan area in Lao PDR (reference 1 and internal reports).
   * Retrospective approach: To determine COVID-19 circulation within the cohort before the appearance of the first positive cases in December 2019 in Wuhan, China, by retrospective SARS-CoV-2 RNA detection in samples collected from a cohort of 1092 households, including 5400 study participants, followed-up between March 2015 and February 2019 (LACORIS project) (1 and internal reports).
   * Prospective approach: To determine COVID-19 progression, over a one-year period from the beginning of the project, by SARS-CoV-2 RNA detection in individuals expressing an influenza-like illness.
   * For this, intra-familial and intra-community transmission rate and context will be evaluated by SARS-CoV-2 RNA detection in contacts of COVID-19 positive cases detected during the prospective phase of the project.
   * To assess past SARS-CoV-2 circulation by screening specific antibodies from saliva swabs in a randomized group of the cohort study.

   In animals:

   - To investigate SARS-CoV-2 transmission to pets and domestic animals by RNA detection in animals living with or near positive cases detected during the prospective phase of the project.
4. STUDY SITES AND POPULATION

   The study will cover 1092 households, including 5400 study participants living in 25 villages within the administrative boundaries of the Vientiane metropolitan area. A household was defined as a group of individuals living on the same plot of land (one or more houses) or in the same building (apartment) and sharing their meals All study co-investigators will be trained before the beginning and during the study on the specific aspects of the study.
5. RESEARCH FLOWCHART

5.1 Flowchart of the participant with ILI symptoms

All family members more than 6 months living with SARS-CoV-2 positive individuals will have non-invasive exam for SARS-CoV-2 detection (nasal, throat, swab, saliva) and a questionnaire.

Participation in the study

Information: All participants will be handed a written information form to participate in the research. This form will provide information on the scope and intent of the study as well as the obligations of the study investigators and expectations from cohort members.

Collection of consent: Before the beginning of the study, an appointment with the investigative surveillance team at the household will be scheduled to explain the details of the project. These details include taking respiratory swab samples in case of influenza-like disease for the patient and family members. The team will hand in the information form and will collect the written consent form from each willing household member, previously signed by three people (Interviewer, parent or guardian, witness/family member)

Cohort participation:

The project study will extend over a year period and will begin as soon as the ethical clearance will be obtained. Households will be selected from household registries and will be enrolled into the cohort via door-to-door sampling, according to the database already set up at CILM. A household is defined as a group of individuals living on the same plot of land (one or more houses) or in the same building (apartment) and sharing meals. Over a year, active case finding for influenza-like illness (ILI) will be conducted among the cohort through weekly phone calls (N=500) to each household by staff at CILM. To increase the likelihood of pathogen identification, study participants will be encouraged to self-report occurrence of symptoms to allow early collection of specimens. As soon as a case meets the ILI-WHO criteria, a free of charge visit will be organised on the same day by the field-trained healthcare staff (the investigative surveillance team) to interview and verify the disease eligibility criteria, to complete a disease investigation questionnaire, where details about the symptomatology will be collected.

Diagnosis results and ILI Follow-up:

The results of COVID 19 analysis (positive or negative) will be transmitted to the NCLE (National Center for Laboratory and Epidemiology).

If the result is COVID19 positive, the NCLE will send it to the "National Taskforce Committee for prevention, control and response COVID-19 pandemic". The COVID-19 positive patient will be taken care by this national Committee and followed up according to the official procedures.

According to the Committee recommendations, all family members living with the COVID-19 patient will be sampled in order to look for asymptomatic infections. In all other cases (detection of another respiratory virus or negative results), the result will be returned on site, in written form, directly to the participant (adult or children between 12 and 18 years old) or to the parent or the guardian (children under 12 years old or adult with psychiatric disorders) by the interviewer. The participants will be referred to medical doctors or to the local healthcare structures to be treated. There are four general hospitals in Vientiane and several local healthcare structures in each of the 25 villages included in our study. When a patient will develop ILI, the doctor in our team will advise him on any treatment to be taken, on the preventive measures to be taken to avoid contamination of other members of his family and will direct him to the closest healthcare structure. Except in exceptional cases, no logistical (transport) or medical support is recommended in the project.

Patients or their family will be attended 60 days later to determine the overall health status, including hospitalisation or death.

5.2 End of research

At the end of the study, a final report will be communicated to each household and the results will be explained by the interviewer.

Each week, the head of the household will be contacted by phone to ask if one member of his family has developed signs of illness. If there is no news from a participant for 3 consecutive weeks, an investigator will go on site to conduct more precise investigations.

5.3 Questionnaires

Overall, the study includes two kind of questionnaires:

A household enrolment questionnaire, including sociodemographic details. Census questions asked upon enrollment to build a database of participating villages for purposes of weekly home visits, disease investigation, and follow-up investigation. This questionnaire will be filled in by the interviewer for each household, at the time of the enrolment, when the information form will be handed in and the signature of the informed consent will be obtained.

A disease investigation questionnaire, including details of the ILI disease. Questions asked will provide information on the person reporting with illness and include basic clinical observations and other information relevant to understanding the source of the illness. This questionnaire will be filled in by the interviewer at the time of the sample collection.

Specimens to be collected using standard protocols include:

* Upper Respiratory swabs (saliva, throat and nasal swabs): samples will be collected on transport medium according to the recommendations of the "National Taskforce Committee for prevention, control and response COVID-19 pandemic". Each sample will be collected by trained field staff using sterile Nylon swabs with plastic shafts and inserted in the sterile cryovial containing universal transport media (UTM).
* The samples will be placed and transported in refrigerated coolers to CILM for testing.
* The patient identification number (see below) will be linked by a relational database and pre-printed labels placed on the questionnaire and on any specimen collected
* Specific qPCR for SARS-CoV2 (targeting RdRp, N and E genes) as well as Pan-coronavirus targeting RdRp will be performed on RNA extracted from retrospective and prospective nasal swabs, throat swabs, and sputum specimens. The analyses will be performed at CILM (Vientiane, Laos). Each positive sample will be sequenced and compared to reference sequences.
* Specific IgG testing will be performed by luminex and ELISA technologies from saliva swabs.
* After testing, the samples will be stored at -80°C at CILM until further analysis upon request for at least 15 years. The samples could be destroyed after at least 15 years upon request from the authorities of Lao PDR and the staff manager of CILM.
* Upon request from the coordinating investigators of the study (Phimpha Paboriboune and Eric Leroy) and agreement of the scientific committee, genetic materials from positive samples will be sent to MIVEGEC UMR IRD 224-CNRS 5290-Université de Montpellier - IRD (911, avenue Agropolis, 34394 Montpellier France) for further analyses that cannot be performed at CILM or for whole genome sequencing.

ELIGIBILITY:
All permanent residents of the household who meet the inclusion criteria of > 6 months old and living in their respective village for at least 6 months will be eligible to participate. All people from the anterior LACORIS study (2015-2019), will be invited to participate to the study.

Over a year, active case finding for influenza-like illness (ILI) will be conducted among the cohort by staff at CILM. The suspected ILI cases will be first identified using the WHO clinical case definition of ILI and Covid 19 as either with:

Acute onset of fever (> 37.5˚C axillary temperature or > 38˚C tympanic temperature) AND cough; OR Acute onset of ANY ONE OR MORE of the following signs or symptoms: Fever, cough, general weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnoea, anosmia (loss of smell) or ageusia (loss of taste).

with symptoms with onset within the last 10 days.

Inclusion Criteria:

* Living in their respective village for 6 months or more.
* Physically reside in the village for more than 80% of the time during the duration of the study.
* Study subjects ≥ 6 months of age (no upper age limit).
* Consent form signed by patient, or if under 18 years of age or patients with learning difficulty or other vulnerability with impaired ability to decide on consent, signed by parent or guardian.
* Agrees to comply with study requirements.

Exclusion Criteria:

* Study subjects under the age of 6 months.
* Study subjects or parents/guardians that do not accept participation.
* Study subjects or parents/guardians who refuse to sign informed consent.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will cover 1092 households, including 5400 study participants living in 25 villages within the administrative boundaries of the Vientiane metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 RNA in respiratory samples collected from influenza-like illness patients from cohort study 2020-2021 | Months 12
  Number of participants SARS-CoV-2 positive among total number of participants tested

SECONDARY OUTCOMES:
Prevalence of SARS-CoV-2 RNA in respiratory samples from influenza-like illness patients from cohort study between 2015 and 2019 | Months 12
  Number of respiratory samples positive for SARS-CoV-2 over the total number of respiratory samples from the 2015-2019 cohort

OTHER OUTCOMES:
Prevalence of SARS-CoV-2 RNA in respiratory samples from intrafamilial contacts of influenza-like illness patients (2020-2021) | Months 12
  Number of SARS-CoV-2 positive samples among the total number of samples collected from participants living within the family nucleus of influenza-like illness patients
Prevalence of SARS-CoV-2 IgG among 1000 individuals randomly selected from the 2020-2121 study cohort. IgG will be assayed in saliva samples | Months 12
  Number of participants IgG positive over a thousand, randomly selected, participants tested.
Prevalence of SARS-CoV-2 RNA in respiratory and faecal samples collected from companion animals living with influenza-like illness patients | Months 12
  Number of pet animals positive for SARS-CoV-2 over the total number of pets tested

CONTACTS AND LOCATIONS:
Overall Officials: Phimpha PABORIBOUNE, MD, PhD, Principal Investigator — Centre d'Infectiologie Lao-Christophe Mérieux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudge JW, Inthalaphone N, Pavlicek R, Paboriboune P, Flaissier B, Monidarin C, Steenkeste N, Davong V, Vongsouvath M, Bonath KA, Messaoudi M, Saadatian-Elahi M, Newton P, Endtz H, Dance D, Paranhos Baccala G, Sanchez Picot V. "Epidemiology and aetiology of influenza-like illness among households in metropolitan Vientiane, Lao PDR": A prospective, community-based cohort study. PLoS One. 2019 Apr 5;14(4):e0214207. doi: 10.1371/journal.pone.0214207. eCollection 2019. PMID 30951544
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Zhang T, Wu Q, Zhang Z. Probable Pangolin Origin of SARS-CoV-2 Associated with the COVID-19 Outbreak. Curr Biol. 2020 Apr 6;30(7):1346-1351.e2. doi: 10.1016/j.cub.2020.03.022. Epub 2020 Mar 19. PMID 32197085
- [Background] Lam TT, Jia N, Zhang YW, Shum MH, Jiang JF, Zhu HC, Tong YG, Shi YX, Ni XB, Liao YS, Li WJ, Jiang BG, Wei W, Yuan TT, Zheng K, Cui XM, Li J, Pei GQ, Qiang X, Cheung WY, Li LF, Sun FF, Qin S, Huang JC, Leung GM, Holmes EC, Hu YL, Guan Y, Cao WC. Identifying SARS-CoV-2-related coronaviruses in Malayan pangolins. Nature. 2020 Jul;583(7815):282-285. doi: 10.1038/s41586-020-2169-0. Epub 2020 Mar 26. PMID 32218527
- [Background] Li W, Shi Z, Yu M, Ren W, Smith C, Epstein JH, Wang H, Crameri G, Hu Z, Zhang H, Zhang J, McEachern J, Field H, Daszak P, Eaton BT, Zhang S, Wang LF. Bats are natural reservoirs of SARS-like coronaviruses. Science. 2005 Oct 28;310(5748):676-9. doi: 10.1126/science.1118391. Epub 2005 Sep 29. PMID 16195424
- [Background] Ar Gouilh M, Puechmaille SJ, Diancourt L, Vandenbogaert M, Serra-Cobo J, Lopez Roig M, Brown P, Moutou F, Caro V, Vabret A, Manuguerra JC; EPICOREM consortium. SARS-CoV related Betacoronavirus and diverse Alphacoronavirus members found in western old-world. Virology. 2018 Apr;517:88-97. doi: 10.1016/j.virol.2018.01.014. Epub 2018 Feb 23. PMID 29482919
- [Background] Leroy EM, Ar Gouilh M, Brugere-Picoux J. The risk of SARS-CoV-2 transmission to pets and other wild and domestic animals strongly mandates a one-health strategy to control the COVID-19 pandemic. One Health. 2020 Dec;10:100133. doi: 10.1016/j.onehlt.2020.100133. Epub 2020 Apr 13. No abstract available. PMID 32363229
- [Background] Shi J, Wen Z, Zhong G, Yang H, Wang C, Huang B, Liu R, He X, Shuai L, Sun Z, Zhao Y, Liu P, Liang L, Cui P, Wang J, Zhang X, Guan Y, Tan W, Wu G, Chen H, Bu Z. Susceptibility of ferrets, cats, dogs, and other domesticated animals to SARS-coronavirus 2. Science. 2020 May 29;368(6494):1016-1020. doi: 10.1126/science.abb7015. Epub 2020 Apr 8. PMID 32269068
- [Background] Gouilh MA, Puechmaille SJ, Gonzalez JP, Teeling E, Kittayapong P, Manuguerra JC. SARS-Coronavirus ancestor's foot-prints in South-East Asian bat colonies and the refuge theory. Infect Genet Evol. 2011 Oct;11(7):1690-702. doi: 10.1016/j.meegid.2011.06.021. Epub 2011 Jul 8. PMID 21763784
- [Background] Lacroix A, Duong V, Hul V, San S, Davun H, Omaliss K, Chea S, Hassanin A, Theppangna W, Silithammavong S, Khammavong K, Singhalath S, Greatorex Z, Fine AE, Goldstein T, Olson S, Joly DO, Keatts L, Dussart P, Afelt A, Frutos R, Buchy P. Genetic diversity of coronaviruses in bats in Lao PDR and Cambodia. Infect Genet Evol. 2017 Mar;48:10-18. doi: 10.1016/j.meegid.2016.11.029. Epub 2016 Dec 6. PMID 27932284
- [Background] Afelt A, Lacroix A, Zawadzka-Pawlewska U, Pokojski W, Buchy P, Frutos R. Distribution of bat-borne viruses and environment patterns. Infect Genet Evol. 2018 Mar;58:181-191. doi: 10.1016/j.meegid.2017.12.009. Epub 2017 Dec 23. PMID 29277555
- [Background] Greatorex ZF, Olson SH, Singhalath S, Silithammavong S, Khammavong K, Fine AE, Weisman W, Douangngeun B, Theppangna W, Keatts L, Gilbert M, Karesh WB, Hansel T, Zimicki S, O'Rourke K, Joly DO, Mazet JA. Wildlife Trade and Human Health in Lao PDR: An Assessment of the Zoonotic Disease Risk in Markets. PLoS One. 2016 Mar 23;11(3):e0150666. doi: 10.1371/journal.pone.0150666. eCollection 2016. PMID 27008628
- [Background] Ceron JJ, Lamy E, Martinez-Subiela S, Lopez-Jornet P, Capela E Silva F, Eckersall PD, Tvarijonaviciute A. Use of Saliva for Diagnosis and Monitoring the SARS-CoV-2: A General Perspective. J Clin Med. 2020 May 15;9(5):1491. doi: 10.3390/jcm9051491. PMID 32429101
- [Background] Randad PR, Pisanic N, Kruczynski K, Manabe YC, Thomas D, Pekosz A, Klein SL, Betenbaugh MJ, Clarke WA, Laeyendecker O, Caturegli PP, Larman HB, Detrick B, Fairley JK, Sherman AC, Rouphael N, Edupuganti S, Granger DA, Granger SW, Collins M, Heaney CD. COVID-19 serology at population scale: SARS-CoV-2-specific antibody responses in saliva. medRxiv [Preprint]. 2020 May 26:2020.05.24.20112300. doi: 10.1101/2020.05.24.20112300. PMID 32511537
- [Background] Faustini SE, Jossi SE, Perez-Toledo M, Shields AM, Allen JD, Watanabe Y, Newby ML, Cook A, Willcox CR, Salim M, Goodall M, Heaney JL, Marcial-Juarez E, Morley GL, Torlinska B, Wraith DC, Veenith TV, Harding S, Jolles S, Ponsford MJ, Plant T, Huissoon A, O'Shea MK, Willcox BE, Drayson MT, Crispin M, Cunningham AF, Richter AG. Detection of antibodies to the SARS-CoV-2 spike glycoprotein in both serum and saliva enhances detection of infection. medRxiv [Preprint]. 2020 Jun 18:2020.06.16.20133025. doi: 10.1101/2020.06.16.20133025. PMID 32588002